CLINICAL TRIAL: NCT03470324
Title: Combined Stimulation of Subthalamic Nucleus and Substantia Nigra Pars Reticulata for Dysphagia: A Randomized Controlled Multicenter Trial
Brief Title: Combined Stimulation of STN and SNr for Dysphagia in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Daniel Weiss, Clinical Professor, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 686/2017BO1
Record Dates: First submitted 2017-12-30; First posted 2018-03-19 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Parkinson's Disease; Dysphagia
Keywords: Parkinson's disease; Dysphagia; Parkinsonian Disorders; Neurodegenerative Diseases; Movement Disorders; Nervous System Diseases; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Deep brain stimulation; substantia nigra pars reticulata; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Parkinsonian Disorders; Neurodegenerative Diseases; Movement Disorders; Nervous System Diseases; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [standard STN] + swallowing therapy (Active Comparator): standard stimulation on subthalamic (STN) contacts plus swallowing therapy
  Interventions: Device: [standard STN]; Behavioral: Swallowing therapy
- [STN+SNr] + swallowing therapy (Experimental): Combined stimulation of the subthalamic nucleus (STN) and the substantia nigra pars reticulata (SNr) plus swallowing therapy
  Interventions: Device: [STN+SNr]; Behavioral: Swallowing therapy

INTERVENTIONS:
Device: [standard STN] — standard stimulation on subthalamic (STN) contacts High frequency deep brain stimulation with variable (best individual) stimulation on subthalamic contacts
  Other Names: subthalamic deep brain stimulation
  Arms: [standard STN] + swallowing therapy
Device: [STN+SNr] — Combined stimulation of the subthalamic nucleus (STN) and the substantia nigra pars reticulata (SNr) high frequency deep brain stimulation of combined (best individual) subthalamic and nigral stimulation
  Other Names: combined subthalamic and nigral stimulation
  Arms: [STN+SNr] + swallowing therapy
Behavioral: Swallowing therapy — Swallowing therapy with speech therapist

SUMMARY:
20 patients with idiopathic Parkinson's disease and dysphagia will be included into this randomised controlled double-blinded parallel group clinical trial. The treatment consists of two different stimulation settings using (i) conventional stimulation of the subthalamic nucleus [standard STN] as active comparator and (ii) combined stimulation of active electrode contacts located in both the subthalamic nucleus and substantia nigra pars reticulata [STN+SNr]. Both groups receive additional swallowing therapy as standard of care.

DETAILED DESCRIPTION:
The primary endpoint of this study is to investigate the efficacy and safety of combined [STN+SNr] stimulation by "interleaving stimulation" as compared to [standardSTN] after 8 weeks on dysphagia. The Trial is designed as superiority study with an 81% power to detect a clinically relevant mean improvement of 2 points on the Penetration Aspiration Scale for fluids (two-tailed p < 0.05). To this end 20 patients will be randomized. After a common baseline assessment in [standardSTN], patients will be randomized to either [standardSTN] or [STN+SNr] in 1:1 ratio (10 per arm). The primary endpoint assessment is scheduled 8 weeks from baseline assessment (V2). Both treatment arms will receive swallowing therapy as standard of care.

The rationale for this study comes from the association of swallowing and oral transport to neuronal integration upon the substantial nigra pars reticulate (SNr)-superior colliculus (SC) pathway (Rossi et al., 2016). Deep brain stimulation of the SNr has been put forward to modulate brainstem circuitry through its monosynaptic brainstem projections to the SC and to the pedunculopontine nucleus (PPN) (Chastan et al., 2009, Weiss et al., 2013, Rossi et al., 2016).

Secondary outcome measures include anamnestic assessments on dysphagia, clinical global impression, freezing of gait and falls, balance, quality of life, neuropsychiatric symptoms and suicidality. Secondary outcome measures also include clinical assessment of dysphagia (Site of Swallow Reflex Initiation, Test of Mastication and Swallowing solids, pharyngeal residue) as well as motor symptoms with MDS-UPDRS III, Capsit-PD and Freezing of Gait Assessment Course.

ELIGIBILITY:
Inclusion Criteria:

* cognitive competence to consent
* Idiopathic Parkinson's disease (according to the "British Brain Bank criteria" (Hughes, 1992) including genetic forms
* Therapy with STN-DBS (deep brain stimulation) (ACTIVA pulse generators) at least six months from surgery
* Activa PC (Primary Cell) or Activa RC (Rechargeable Cell) as implanted pulse generator with "Interleaving" programming option
* Localization of an active electrode contact in the sub thalamic nucleus
* Localization of the caudal electrode contacts in the substantia nigra pars reticulata area (coordinates relative to midcommisural Point (MCP): left: -7mm ≤ x ≤ -12mm; -2mm ≤ y ≤ -6mm; -6mm ≤ z ≤ -10mm right: 7mm ≤ x ≤ 12mm; -2mm ≤ y ≤ -6mm; -6mm ≤ z ≤ -10mm (x = medio-lateral, y = anterio-posterior, z = rostro-caudal)
* ≥ 30% improvement in UPDRS III with 'standard STN' compared to 'stimulation off' in dopaminergic off
* Penetration-Aspiration-Scale ≥ 3 or more than 20% utilization of vallecular space and/or pyriform sinuses post swallowing
* Disease duration ≥ 5 years
* Age: between 18 and 80 years
* Dopaminergic medication constant for at least two weeks prior to study enrollment
* Written informed consent

Exclusion Criteria:

* Participation in other clinical trials within the past three months and during study enrolment
* Cognitive impairment (Mini Mental State Exam < 20)
* Severe depressive episode with or without psychotic symptoms and suicidality (ICD-10: F32.2, F32.3), psychosis (ICD-10: F23.-)
* Other severe pathological chronic condition that might confound treatment effects or interpretation of the data
* Pregnancy
* Infection and pneumonia at the time of study enrollment
* Other competing cause for dysphagia (e.g. stroke, operation, radiotherapy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Outcome after eight weeks (V2) with reference to baseline (V1)
  8-point interval scale (range 1 - 8) to describe penetration and aspiration events . Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. (Rosenbek et al, 1996). The score is obtained in swallowing of fluids

SECONDARY OUTCOMES:
MDS-UPDRS parts I, II, III and IV | Outcome after eight weeks (V2) with reference to baseline (V1)
  Rating Scale for symptoms of Parkinson's Disease: I Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications.
Capsit-PD | Outcome after eight weeks (V2) with reference to baseline (V1)
  Walking distance of 7m. Patient has to walk that distance back and forth. The time is measured as well as the number of steps needed for each way. Also, freezing episodes are counted.
Freezing of Gait Assessment Course (FOG-AC) | Outcome after eight weeks (V2) with reference to baseline (V1)
  Patients were asked to sit down on a chair, then stand up and walk to a floor mark .Within the mark they performed two 360° turns, clockwise (cw) and counter-clockwise (ccw). Then: open and walk through the door, turn outside, and come back to their chair.
  Four situations were rated: The start to walk, the turning (cw and ccw), and the passing through the door. 0 points: no festination and no FOG , 1 point: festination or any hastening steps. 2 points: FOG (trembling-in-place or total akinesia), which the patient could overcome himself. 3points: abortion of the task or need of interference by the examiner. Three levels of multiple tasking were applied: First passage;: no additional task ("walking"). Second passage: carrying a tray with a plastic cup full of water. Third passage: motor task and a mental task ("carrying and calculation"). (Ziegler et al. 2010)
PDQ-39 | Outcome after eight weeks (V2) with reference to baseline (V1)
  The 39-item Parkinson's Disease Questionnaire is a widely used patient-reported clinical trial endpoint, where patients are asked about their health-related quality of life related to Parkinson's disease.
Dysphagia-related Quality of Life (SWAL-QoL) | Outcome after eight weeks (V2) with reference to baseline (V1)
  48-item quality-of-life outcomes tool for dysphagia researchers and clinicians
Clinical global impression self | Outcome after eight weeks (V2)
  (self-reporting, caregiver-reporting)
Diary on swallowing an related complications | Outcome after eight weeks (V2) with reference to baseline (V1)
  complications (cough, suffocation, bronchitis, aspiration pneumonia)
Site of Swallow reflex initiation | Outcome after eight weeks (V2) with reference to baseline (V1)
  Two FEES outcome variables-delayed initiation of the pharyngeal reflex and postswallow pyriform sinus pooling(Scott et al 1998)
Test of Mastication and Swallowing solids (TOMASS) | Outcome after eight weeks (V2) with reference to baseline (V1)
  The Test of Masticating and Swallowing Solids (TOMASS) was developed as a quantitative assessment of solid bolus ingestion. For each study the test required participants to ingest a commercially available cracker with instructions to 'eat this as quickly as is comfortably possible'. Further averaged measures were derived including the number of masticatory cycles and swallows per bite, and time per bite, masticatory cycle and swallow.
Pharyngeal Residue Visual Analogue Scale (VAS) | Outcome after eight weeks (V2) with reference to baseline (V1)
  With FEES the pharyngeal residue (Sinus piriformis and vallecular) are rated on a visual analogue scale
Functional oral intake scale (FOIS) | Outcome after eight weeks (V2) with reference to baseline (V1)
  Scale to assess oral intake (7 points indicate full oral intake without restrictions, 1 points indicates no oral intake possible, 1-3 tube dependent) (Crary et al. 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tübingen, Tübingen, Germany

REFERENCES:
- [Background] Weiss D, Walach M, Meisner C, Fritz M, Scholten M, Breit S, Plewnia C, Bender B, Gharabaghi A, Wachter T, Kruger R. Nigral stimulation for resistant axial motor impairment in Parkinson's disease? A randomized controlled trial. Brain. 2013 Jul;136(Pt 7):2098-108. doi: 10.1093/brain/awt122. Epub 2013 Jun 11. PMID 23757762
- [Background] Rossi MA, Li HE, Lu D, Kim IH, Bartholomew RA, Gaidis E, Barter JW, Kim N, Cai MT, Soderling SH, Yin HH. A GABAergic nigrotectal pathway for coordination of drinking behavior. Nat Neurosci. 2016 May;19(5):742-748. doi: 10.1038/nn.4285. Epub 2016 Apr 4. PMID 27043290
- [Background] Chastan N, Westby GW, Yelnik J, Bardinet E, Do MC, Agid Y, Welter ML. Effects of nigral stimulation on locomotion and postural stability in patients with Parkinson's disease. Brain. 2009 Jan;132(Pt 1):172-84. doi: 10.1093/brain/awn294. Epub 2008 Nov 11. PMID 19001482
- [Background] Scholten M, Klemt J, Heilbronn M, Plewnia C, Bloem BR, Bunjes F, Kruger R, Gharabaghi A, Weiss D. Effects of Subthalamic and Nigral Stimulation on Gait Kinematics in Parkinson's Disease. Front Neurol. 2017 Oct 17;8:543. doi: 10.3389/fneur.2017.00543. eCollection 2017. PMID 29089922
- [Background] Hidding U, Gulberti A, Horn A, Buhmann C, Hamel W, Koeppen JA, Westphal M, Engel AK, Gerloff C, Weiss D, Moll CK, Potter-Nerger M. Impact of Combined Subthalamic Nucleus and Substantia Nigra Stimulation on Neuropsychiatric Symptoms in Parkinson's Disease Patients. Parkinsons Dis. 2017;2017:7306192. doi: 10.1155/2017/7306192. Epub 2017 Jan 26. PMID 28246572
- [Background] Weiss D, Breit S, Wachter T, Plewnia C, Gharabaghi A, Kruger R. Combined stimulation of the substantia nigra pars reticulata and the subthalamic nucleus is effective in hypokinetic gait disturbance in Parkinson's disease. J Neurol. 2011 Jun;258(6):1183-5. doi: 10.1007/s00415-011-5906-3. Epub 2011 Feb 2. No abstract available. PMID 21287187